CLINICAL TRIAL: NCT06915766
Title: Intermediate-Size Patient Population Expanded Access to Bezuclastinib for Patients With NonAdvanced Systemic Mastocytosis or Advanced Systemic Mastocytosis
Brief Title: Expanded Access to Bezuclastinib for Patients With NonAdvanced Systemic Mastocytosis or Advanced Systemic Mastocytosis
Status: Available | Type: Expanded Access
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CGT9486-IEAP-001
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Systemic Mastocytoses, Indolent; Systemic Mastocytoses, Aggressive
Keywords: Systemic Mastocytosis; NonAdvanced Systemic Mastocytosis; Advanced Systemic Mastocytosis; Systemic Mastocytosis with an associated hematologic neoplasm (SM-AHN); Aggressive Systemic Mastocytosis (ASM); Mast Cell Leukemia (MCL); Bone Marrow Mastocytosis (BMM)
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Bezuclastinib — Drug: Bezuclastinib Tablets
  Other Names: CGT9486

SUMMARY:
The purpose of this expanded access program (EAP) protocol is to provide investigational bezuclastinib to patients with a diagnosis of nonadvanced systemic mastocytosis (NonAdvSM) or advanced systemic mastocytosis (AdvSM) who have received and failed or been intolerant to at least one standard approved therapy and/or have no comparable or satisfactory alternative therapy options.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to provide written informed consent and commit to EAP assessments.
* ≥18 years of age.
* Able to swallow tablets.
* Diagnosed with ASM, SM-AHN, MCL, BMM, ISM, or SSM according to the 2022 WHO Classification for SM
* Not receiving adequate disease control on current therapy(ies).
* Have clinically acceptable laboratory screening results.

Exclusion Criteria:

* Patients who are eligible for and/or enrolled in an on-going bezuclastinib clinical trial.
* Patients who discontinued investigational use of bezuclastinib in previous clinical trials due to toxicity or withdrawal of consent.
* Pregnant or currently breastfeeding.
* Prior or ongoing clinically significant illness or medical or physical condition

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Easton, MD, PhD, Study Director — Cogent Biosciences, Inc.
Locations (17):
- United States (17):
  - Orso Health/Modena Asthma Allergy, La Jolla, California
  - Scripps Green Hospital, La Jolla, California
  - Sneeze Wheeze & Itch Associates LLC Clinical Research Center, Normal, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Walter Reed, Bethesda, Maryland
  - AllerVie Health, Glenn Dale, Maryland
  - Boston Specialists, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Michigan Medicine- University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Blood Cancer Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - AIR Care, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas